CLINICAL TRIAL: NCT04459260
Title: Treating Perfectionism Using Internet-Based Cognitive Behavior Therapy: A Randomized Controlled Trial Comparing Cognitive Behavior Therapy to Unified Protocol
Brief Title: Treating Perfectionism Using Internet-Based Cognitive Behavior Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Uppsala University (Other); Linkoeping University (Other Government); Stockholm University (Other); University College, London (Other)
Responsible Party: Principal Investigator, Alexander Rozental, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UU2020-0001
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Perfectionism; Anxiety; Depression; Stress
Keywords: Perfectionism; Cognitive Behavior Therapy; Unified Protocol; Internet-based; Randomized controlled trial
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavior Therapy (Experimental): An eight-week Internet-based self-guided treatment, delivered with guidance on demand from therapists in training. The treatment is based on cognitive behavior therapy and includes both cognitive interventions, e.g., cognitive restructuring and behavioral experiments, and behavioral interventions, behavioral activation. The treatment was manualized by Egan et al. (2016) and has been tested in several clinical trials, both via the Internet and face-to-face.
  Interventions: Behavioral: Cognitive Behavior Therapy
- Unified Protocol (Active Comparator): An eight-week Internet-based self-guided treatment, delivered with guidance on demand from therapists in training. The treatment is based on a transdiagnostic approach derived from cognitive behavior therapy called Unified Protocol, focusing on the shared emotional aspects underlying depression and anxiety disorders. The treatment was manualized by Ellard et al. (2010) and has been tested in several clinical trials, but so far not over the Internet.
  Interventions: Behavioral: Unified Protocol

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy — A standardized evidence-based treatment manual based on cognitive behavior therapy, developed specifically for targeting perfectionism (Egan et al., 2016). Includes the following components: 1) providing psychoeducation about perfectionism and creating an individualized conceptualization 2) broadening the domains for self-evaluation 3) testing out beliefs and predictions, and 4) addressing personal standards and self-criticism.
  Week 1: Understanding your perfectionism.
  Week 2: Your own model, values, and motivation.
  Week 3: Surveys and experiments.
  Week 4: Dealing with perfectionistic behaviors.
  Week 5: New ways of thinking.
  Week 6: Self-criticism and self-compassion.
  Week 7: Self-worth.
  Week 8: Maintain and continue positive change.
  Arms: Cognitive Behavior Therapy
Behavioral: Unified Protocol — A standardized evidence-based treatment manual based on cognitive behavior therapy, developed to target the shared emotional factors in depression and anxiety disorders (Ellard et al., 2010). Fundamental to this approach is to register and become more aware of the emotions, cognitions, and physical sensations that occur in difficult situation, and to try out more adaptive ways of coping in these instances.
  Week 1: Emotional symptoms.
  Week 2: Understanding your emotions.
  Week 3: Emotional awareness.
  Week 4: Thoughts.
  Week 5: Behaviors.
  Week 6: Emotional exposure.
  Week 7: Continued emotional exposure.
  Week 8: Planning ahead.
  Arms: Unified Protocol

SUMMARY:
Perfectionism is characterized by setting high standards and striving for achievement, sometimes at the expense of social relationships and wellbeing. Despite sometimes being viewed as a positive feature by others, people with perfectionism tend to be overly concerned about their performance and how they are being perceived by people around them. This tends to create inflexible standards, cognitive biases, and performance-related behaviors that maintain a belief that self-worth is linked to accomplishments. Cognitive behavior therapy has been shown to be a viable treatment for perfectionism, both in terms of reducing levels of perfectionism and improving psychiatric symptoms. Furthermore, a number of recent studies indicate that it can be successfully delivered via the Internet, both with regular support and guidance on demand from a therapist. In the present study protocol, a clinical trial for perfectionism is described and outlined. In total, 128 participants will be recruited and randomized to either a treatment that has already been demonstrated to have many benefits, Internet-based Cognitive Behavior Therapy for perfectionism (iCBT-P), or an active comparison condition, Internet-based Unified Protocol (iUP), targeting the emotions underlying depression and anxiety disorders. The results will be investigated with regard to self-reported outcomes of perfectionism, psychiatric symptoms, self-compassion, and quality of life, at post-treatment and at six- and 12-month follow-up. Both iCBT-P and iUP are expected to have positive effects, but the difference between conditions and adherence to respective treatment are currently unknown and will be explored. The clinical trial is believed to lead to a better understanding of how perfectionism can be treated, with the aim of providing efficacious treatments in an accessible format via the Internet.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years
* Adequate reading and writing levels in Swedish
* A computer, smartphone, or tablet with Internet access
* Elevated levels of perfectionism, as determined by a score of >29 on the subscale Concerns over Mistakes on the Frost Multidimensional Perfectionism Scale

Exclusion Criteria:

* Diagnoses warranting immediate care, e.g., anorexia nervosa, substance abuse, bipolar disorder, psychosis, and schizophrenia
* Severe depression, as determined by a score of >15 points on the Patient Health Questionnaire - 9 Items
* Suicidality, as determined by >2 points on the item on suicidal ideation on the Patient Health Questionnaire - 9 Items

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Clinical Perfectionism Questionnaire (CPQ) | One month
  The CPQ is a self-report measure determining the level of perfectionism and consists of 12 items that are scored on a four-point Likert-scale 1-4 ("Not at all" to "All of the time"), with two items that are in reverse (items 2 and 8), and employing a time-frame of one month to increase its clinical usefulness. The CPQ was translated to Swedish in a previous clinical trial, demonstrating good convergent and discriminant validity when compared to self-report measures of perfectionism and psychiatric symptoms, as well as adequate internal consistency and test-retest reliability (McMahan et al., submitted).
Frost Multidimensional Perfectionism Scale (FMPS) | One month
  The FMPS is self-report measure determining the level of perfectionism and is scored on a five-point Likert-scale 1-5 ("Strongly disagree" to "Strongly agree"), with a total of 35 items that cover the six separate subscales Concern over Mistakes, Personal Standards, Doubts about Action, Parental Expectations, Parental Criticism, and Organization. However, only the two first are usually of interest in clinical trials as the other subscales are considered less related to the two higher-order dimensions of perfectionism (Limburg et al., 2017). The subscales of the FMPS has adequate to excellent internal consistencies and exhibits convergent and discriminant validity when compared to self-report measures of perfectionism and psychiatric symptoms (Purdon, Antony, & Swinson, 1999). The FMPS was originally translated to Swedish by Lundh, Broman, Hetta, and Saboonchi (1994).

SECONDARY OUTCOMES:
Patient Health Questionnaire - 9 Items (PHQ-9) | Two weeks
  The nine-item PHQ-9 assesses the degree of depression and is scored on a four-point Likert-scale 0-3 ("Not at all" to "Nearly every day"). The PHQ-9 is often used as a screening tool for depressive symptoms, has been validated against other self-report measures and clinical interviews of depression, and has an excellent internal consistency (Kroenke et al., 2001).
Generalized Anxiety Disorder - 7 Items (GAD-7) | Two weeks
  The seven-item Generalized Anxiety Disorder (GAD-7) determines the level of anxiety and is scored on a four-point Likert-scale 0-3 ("Not at all" to "Nearly every day"). The GAD-7 is often used for screening for symptoms of anxiety and worry, corresponds well with other similar self-report measures, and has exhibited excellent internal consistency (Spitzer, Kroenke, Williams, & Lowe, 2006).
Brunnsviken Brief Quality of Life (BBQ) | One month
  The 12-item Brunnsviken Brief Quality of Life (BBQ) explores the quality of life in six areas, e.g., leisure and learning, and level of importance, e.g., "my leisure time is important to me", which are then multiplied with each other. The BBQ is scored on a four-point scale 1-4 ("Strongly disagree" to "Strongly agree"), with a range in scores of 0-96. The BBQ demonstrates good convergent and discriminant validity, good classification ability, and has an adequate internal consistency (Lindner et al., 2016).
Self-Compassion Scale - Short Form (SCS-SF) | One month
  The 12-item Self-Compassion Scale - Short Form (SCS-SF) tests the degree of self-compassion and is scored on a five-point scale 1-5 ("Almost never" to "Almost all of the time"). The SCS-SF has been shown to correlate with self-report measures of psychiatric symptoms, and has a good internal consistency (Raes, Pommier, Neff, & Van Gucht, 2011).
Pure Procrastination Scale (PPS) | One month
  The 12-item Pure Procrastination Scale (PPS) determines the level of procrastination and is scored on a five-point Likert-scale 1-5 ("Seldom, or do not agree" to "Very often, or totally agree). The PPS has been shown to have good convergent and discriminant validity, and internal consistency (Rozental, Forsell, et al., 2014; Steel, 2010).
Perceived Stress Scale (PSS) | One month
  The 14-item Perceived Stress Scale (PSS) evaluates the subjective experience of general stress in various situations and is scored on a five-point Likert-scale 0-4 ("Never" to "Very often"), with seven items being scored in reverse (items 4-7, 9-10, and 13). The PSS has been shown to have adequate internal consistency as well as good convergent and discriminant validity (Cohen, Kamarck, & Mermelstein, 1983).
Negative Effects Questionnaire (NEQ) | One month
  Negative Effects Questionnaire (NEQ) will be used to probe for unwanted and adverse events that might arise during treatment, which is scored on a five-point Likert-scale 0-4 ("Not at all" to "Extreme"), and classifies the incidents as caused by the treatment or other circumstances. The NEQ has demonstrated excellent internal consistency and is mainly used to descriptively determine the occurrence and nature of possible negative effects (Rozental, Kottorp, Boettcher, Andersson, & Carlbring, 2016).
Credibility/Expectancy Questionnaire | Two weeks
  The perceived integrity of treatment will be explored using the five-item Credibility/Expectancy Questionnaire (Borkovec & Nau, 1972), which is scored on a 10-point Likert-scale 0-10 (e.g., "Not at all logical" to " Very logical"). It has exhibited good internal consistency and test-retest reliability, with the factor expectancy being correlated with outcomes of treatment (Devilly & Borkovec, 2000).
Domains | One month
  The effects of treatment will be explored using subjective ratings of its impact on different domains. This will entail eight aspects of life that each participant rates on a 10-point Likert-scale 0-10 with regard to how perfectionism is affecting them negatively ("Not at all" to "Very much"): interests/leisure, work/studies, friendships/social life, community engagement/spirituality, family life/parenting, rest/sleep, love/intimate relationships, and physical activity/diet.
Goal attainment | One month
  The effects of treatment will be explored using participants own statements and definitions of their goals of treatment, and to what extent they have lived up to them, rated on a 10-point Likert-scale 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Buhrman, PhD, Principal Investigator — Monica.Buhrman@psyk.uu.se
Locations (1):
- Uppsala University, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No
Masked and anonymised data will be able to retrieve upon request.

REFERENCES:
- [Result] Rozental A, Shafran R, Johansson F, Forsstrom D, Jovicic F, Gelberg O, Molin K, Carlbring P, Andersson G, Buhrman M. Treating perfectionism via the Internet: a randomized controlled trial comparing cognitive behavior therapy to unified protocol. Cogn Behav Ther. 2024 May;53(3):324-350. doi: 10.1080/16506073.2024.2327339. Epub 2024 Mar 14. PMID 38483057
- See also: Study website — https://www.iterapi.se/sites/lizzie/